CLINICAL TRIAL: NCT05692102
Title: Quality of Women Life After Gynacological Malignancies
Brief Title: Quality of Life After Gynacological Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MGAMorsy, principal investigator, Assiut University
Other Study IDs: QOLAGM
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluate quality of life after gynaecological malignancies diagnosis and treatment — diagnosis and treatment

SUMMARY:
Evaluate quality of life after gynaecological malignancies diagnosis and treatment

DETAILED DESCRIPTION:
gynecological cancers represent 10% of new cancer cases among women The main types are cervical, endometrial, ovarian and breast cancers. Each of these is unique in terms of prognosis, treatment, and age at onset.

Early detection and improvement in treatment of these cancers has led to improvements in survival and, consequently, an increase in the number of survivors However, survival is accompanied by several negative aspects, such as fatigue, physical changes, sexual dysfunction, anxiety, and/or depression In addition to the physical and psychological disorders, survivors of gynecological cancer can experience economic problems related to work, or access to loans and insurance Although cancer occurs mainly in older adults, some people, particularly survivors of cervical and ovarian cancer, may experience cancer at an age where work is still of major importance For these women, a return to work represents a return to a normal social life and helps them to regain their self-esteem. Furthermore, work is a source of emotional and financial support and has been shown to enhance health-related quality of life by its positive effect on self-esteem Therefore, special attention must be paid to the well-being of survivors of gynecological cancer, as well as to their social and professional reintegratio is a multidimensional concept which encom passes physical and mental health as well as social well being. Although in recent decades, several studies have focused on and its determinants in survivors of gynecological cancer, has mainly been studied as it pertains to clinical data or with short follow-up durations. Our previous studies in long-term survivors of breast cancer have shown that the likelihood that will depend on other factors increases in line with the length of follow-up since diagnosis.

Due to the improvement in medical science and continuing advancement in early detection and treatment, the expected survival time of cancer patients has become longer. This has resulted in an increased interest in exploring the health-related quality of life of cancer survivors. So, there is a consequent need to satisfy cancer patients' requirements which would enable them to live a healthy life In many cases, cancer patients experience sleep disturbance, depression and poor quality of life after being diagnosed and treated for cancer. So, the assessment of QoL among cancer patients is essential in order to design interventions for improving patients' outcomes Likewise, QoL assessment assists people realize how treatment, disease, and health impact quality of life. Furthermore, it helps to understand potential beneficial and risky aspects of a treatment thus help in weighing the impact of a decision

ELIGIBILITY:
Inclusion Criteria:.patient diagnosed to have gynaecological cancers by histopathology 2.Adult from 20-70 yrs 3. willing and able to participate 4.Early stage 1-2

Exclusion Criteria:

1pre-existing psychological disorders 2.Stage 4 3.severe medical complications as cardiac pt 4.Morbid obesity BMI<40

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible women admitted to Assiut University Women health Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate quality of life after gynaecological malignancies diagnosis and treatment | 2 years
  Evaluate quality of women life after gynaecological malignancies diagnosis and treatment

IPD SHARING:
Plan to Share IPD: Undecided
Evaluate quality of life after gynaecological malignancies diagnosis and treatment